CLINICAL TRIAL: NCT03771326
Title: Preliminary Evidence Suggesting That Acute Administration of KP-10 Induces Insulin Secretion in Normal Weight But Not in Obese Men
Brief Title: KP-10 and Insulin Secretion in Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Quaid-e-Azam University (Other)
Responsible Party: Principal Investigator, Ghulam Nabi, Head of Animal Sciences, Quaid-e-Azam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Kisspeptin12
Record Dates: First submitted 2018-12-04; First posted 2018-12-11 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Kisspeptin Action on Insulin in Healthy Normal Men; Kisspeptin Action on Insulin in Obese Diabetic Men
MeSH Terms: interventions — KISS1 protein, human

STUDY DESIGN:
Intervention Model Description: Fourteen volunteers (aged 20-45 years), including seven adult normal weight healthy men (mean body weight and BMI 75.5±4.8 kg and 23±0.7 kg/m2, respectively) and seven obese men (mean body weight and BMI 115±15 kg and 34±2 kg/m2, respectively), participated in this clinical study
Masking Description: All the individuals were told before the use of Kp-10 administration. however, to avoid psychological effect the exact time was not disclosed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- obese men (Experimental): To the 7 obese men, kisspeptin-10 was intravenously administered (0.5µg/kg BW, prepared under sterile conditions), as a bolus in a volume of 1ml. Blood samples from all the individuals were collected for 30 minutes pre and 120 minutes post-KP-10 administration, at 30 minutes interval. The obtained blood was centrifuged and the plasma insulin was measured by ELISA.
  Interventions: Biological: Kisspeptin-10
- Normal men (Experimental): To the 7 normal BMI mean, kisspeptin-10 was intravenously administered (0.5µg/kg BW, prepared under sterile conditions), as a bolus in a volume of 1ml. Blood samples from all the individuals were collected for 30 minutes pre and 120 minutes post-KP-10 administration, at 30 minutes interval. The obtained blood was centrifuged and the plasma insulin was measured by ELISA.
  Interventions: Biological: Kisspeptin-10

INTERVENTIONS:
Biological: Kisspeptin-10 — Kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany)

SUMMARY:
Induction of insulin secretion by kisspeptin is observed in mouse, pig, rat, and human islets in vitro and in rats, mice and monkeys in vivo, but its mechanism is not fully clear. The present study was designed to investigate the role of KP-10 on insulin secretion in adult healthy and obese men with insulin resistance. The aim of selection of obese persons for the present study was to investigate the effect of acute KP-10 administration in a metabolically challenged condition where the pancreatic beta cells are already highly activated. The long-term objective of this study was to understand the physiological role of kisspeptin signalling in the regulation of insulin secretion in human health and disease.

ELIGIBILITY:
Inclusion Criteria:

* Normal BMI
* Normal renal function
* Normal liver function
* Normal blood count

Exclusion Criteria:

* Disease history
* Diabetes
* Other trauma

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10-29 (Actual); Primary Completion 2013-11-04 (Actual); Study Completion 2014-01-10 (Actual)

PRIMARY OUTCOMES:
Changes in the response of insulin secretion to acute exogenous kisspeptin administration | Each participant was studied up to 4 hours. Blood samples from each individual was collected for 30 minutes pre and 120 minutes post KP-10 administration, at 30 minutes interval.
  The blood samples were obtained and analysed for insulin by Enzyme Linked Immunosorbent Assay to know the differential response of insulin secretion to exogenous kisspeptin-10 administration in healthy and obese men.

IPD SHARING:
Plan to Share IPD: Undecided
This study is already completed. Investigators can disclose participants information after the article is available online.

REFERENCES:
- [Result] Bowe JE, Foot VL, Amiel SA, Huang GC, Lamb MW, Lakey J, Jones PM, Persaud SJ. GPR54 peptide agonists stimulate insulin secretion from murine, porcine and human islets. Islets. 2012 Jan-Feb;4(1):20-3. doi: 10.4161/isl.18261. Epub 2011 Dec 23. PMID 22192948
- [Result] Wahab F, Riaz T, Shahab M. Study on the effect of peripheral kisspeptin administration on basal and glucose-induced insulin secretion under fed and fasting conditions in the adult male rhesus monkey (Macaca mulatta). Horm Metab Res. 2011 Jan;43(1):37-42. doi: 10.1055/s-0030-1268458. Epub 2010 Dec 6. PMID 21136344